CLINICAL TRIAL: NCT00880230
Title: INTENSE: Iliac Artery Treatment With The Invatec Scuba™ Cobalt Chromium Stent
Brief Title: Iliac Artery Treatment With The Invatec Scuba™ Cobalt Chromium Stent (INTENSE)
Acronym: INTENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-999
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Peripheral Artery Disease
Keywords: Iliac Artery Stenting; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Scuba Iliac Stent System (Experimental): Device: Scuba™ iliac stent
  Interventions: Device: Scuba Iliac Stent System

INTERVENTIONS:
Device: Scuba Iliac Stent System — The Scuba™ Stent System consists of a balloon-expandable stent and an over the wire (OTW) delivery system.
  Other Names: Scuba

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Scuba™ stent in subjects with symptomatic claudication or rest pain and angiographic confirmation of de novo or restenotic lesions in the common and/or external iliac artery.

DETAILED DESCRIPTION:
Interventional revascularization strategies for peripheral arterial disease currently available include both surgical and endovascular approaches such as percutaneous transluminal angioplasty (PTA), either as a stand-alone procedure or with the placement of a stent. Cobalt-chromium (CoCr) is an alloy that has been used safely in the manufacture of surgical implants for use in contact with blood, soft tissue and bone for over 10 years. This study will evaluate the SCUBA™ peripheral balloon-expandable cobalt chromium tent system in iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

* Presence of de novo or restenotic lesion(s), located in the common or external iliac artery with ≥50% stenosis
* Subject has lifestyle limiting claudication or rest pain, (Rutherford- Becker scale [clinical category] 2, 3, or 4)
* Target vessel reference diameter is 5mm - 10mm by visual assessment
* Target lesion length < 130mm
* Subject has angiographic evidence of a patent femoral outflow artery in the target limb
* Subject has provided written informed consent
* Subject is able and willing to adhere to required follow-up visits and testing

Exclusion Criteria:

* Subject has lesions in the Common Femoral Artery (CFA), Profundal Femoral Artery (PFA), or Superficial Femoral Artery (SFA) that would require a staged procedure within 30 days of the index procedure (either before or after)
* Target lesion(s) has adjacent, acute thrombus
* Target lesion(s) is highly calcified or was previously treated with a stent
* Subject has a pre-existing target iliac artery aneurysm or perforation or dissection of the target iliac artery
* Subject has an abdominal aortic aneurysm contiguous with the iliac artery target lesion
* Subject has a post-surgical stenosis and anastomotic suture treatments in the native iliac vessel
* Subject has a vascular graft previously implanted in the native iliac vessel
* Subject has tissue loss - Rutherford-Becker clinical category 5 or 6
* History of neutropenia (WBC <3,000/mm3), coagulopathy, or thrombocytopenia (platelet count <80,000/uL)
* International Normalized ratio (INR) greater than 1.5
* Serum creatinine greater than 2.5 mg/dL
* Subject has a known bleeding or hypercoagulability disorder or significant anemia (Hb < 8.0 g/dL) that cannot be corrected
* Subject is participating in an investigational study of a new drug, biologic, or device at the same time of study screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H Gray, DO, Principal Investigator — Greeville Health System; Barry T Katzen, MD, Principal Investigator — Baptist Health South Florida
Locations (3):
- United States (2):
  - Baptist Hospital of Miami, Miami, Florida
  - Greenville Hospital System, Greenville, South Carolina
- Hamburg University Cardiovascular Center, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was for a period of 16 months. Subjects were recruited at medical clinics who participate in clinical trials.
Groups:
- Scuba Iliac Stent System: Device: Scuba Iliac Stent
  Scuba Iliac Stent System: The Scuba Stent System consists of a balloon-expandable stent and an over the wire (OTW) delivery system.
Period: Overall Study
Arm/Group | Scuba Iliac Stent System
Started | 141
Completed | 134
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.90 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 108
Region of Enrollment [Number; unit: participants]
  United States | 59
  Germany | 70
  Switzerland | 12

OUTCOME MEASURES:

1. Primary Outcome: Composite of Major Adverse Events (MAE) Defined as the Occurrence of In-hospital Myocardial Infarction (MI) or Target Segment Revascularization, Target Limb Loss, or Death Within 9 Months Post-procedure.
Description: The analysis is based on the percentage of Intent to Treat subjects (ITT) who experienced the primary endpoint or who had adequate follow-up for the 9-month analysis. A subject had adequate follow-up if he/she had an event or had a follow-up of at least 256 days, allowing for a visit window of 9 months +/- 14 days.
Time Frame: In-hospital and 9 Months
Population: Intent to Treat Population (ITT)
Measure: Number; unit: Percentage of Participants
Groups:
- Scuba Iliac Stent System: Device: Scuba™ iliac stent
  Scuba Iliac Stent System : The Scuba™ Stent System consists of a balloon-expandable stent and an over the wire (OTW) delivery system.
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Participants | 5.2 [2.1 to 10.5]

2. Secondary Outcome: Major Adverse Vascular Events Through 30 Days as a Composite of (MI, Death or Stroke, Stent Thrombosis, Distal Embolization, Arterial Rupture/Perforation, Acute Limb Ischemia, Target Limb Loss, Procedure-related Bleeding Event Requiring Transfusion)
Description: The analysis is based on the number of patients who experienced either an MI, died, had a stroke, stent thrombosis, distal embolization, arterial rupture/perforation limb ischemia, lost a target limb, or had a bleeding event due to the procedure within 30 days after being treated with the Scuba iliac stent.
Time Frame: 30 Days
Population: Intent to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 2.2 [0.5 to 6.2]

3. Secondary Outcome: Device Success
Description: The outcome is based on the successful delivery and deployment of the Scuba iliac stent and the intact retrieval of the delivery system.
Time Frame: At time of deployment
Population: Intent to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 95 [90 to 98]

4. Secondary Outcome: Procedural Success
Description: The outcome is based on the successful delivery and deployment of the Scuba iliac stent and the intact retrieval of the delivery system [Device Success] and the achievement of <30% residual stenosis immediately after stent deployment, without occurrence of in-hospital Major Adverse Events (MAE).
Time Frame: Up to the moment the catheter sheath introducer has been removed
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 86.5 [79.8 to 91.7]

5. Secondary Outcome: Clinical Success
Description: Early Clinical Success (30 days) is defined as improvement of the Rutherford-Becker scale criteria by greater than or equal to one category as obtained at the 30 day follow-up visit.
Time Frame: 30 Days
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 93.8 [88.2 to 97.3]

6. Secondary Outcome: Clinical Success
Description: Late Clinical Success (6 months) is defined as a maintained improvement in Ankle-Brachial Index (ABI) or Thigh-Brachial Index (TBI) assessed as either a) normalized (0.90) or b) an increase by 0.1 from the baseline level and had not decreased by more than 0.15 from the maximum result observed immediately post-procedure. In the absence of ABI/TBI data, Late Clinical Success was assessed in the same manner as Early Clinical Success.
Time Frame: 6 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 69.3 [60 to 77.6]

7. Secondary Outcome: Clinical Success
Description: Late Clinical Success (9 months) is defined as a maintained improvement in Ankle-Brachial Index (ABI) or Thigh-Brachial Index (TBI) assessed as either a) normalized (0.90) or b) an increase by 0.1 from the baseline level and had not decreased by more than 0.15 from the maximum result observed immediately post-procedure. In the absence of ABI/TBI data, Late Clinical Success was assessed in the same manner as Early Clinical Success.
Time Frame: 9 Months
Population: Intent to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 66.4 [57.2 to 74.8]

8. Secondary Outcome: Patency - Primary
Description: Patients were assumed primary patent if the target vessel had continuous flow without revascularization, bypass, or amputation at 6 months.
Time Frame: 6 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 94.9 [89.7 to 97.9]

9. Secondary Outcome: Patency - Primary Assisted
Description: Primary assisted patency is defined as continuous flow assisted with a revascularization when the target vessel has restenosed (0-99%) at any time post-procedure through 6 months.
Time Frame: 6 Months
Population: Intention to Treat (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 1.5 [0.2 to 5.2]

10. Secondary Outcome: Patency - Secondary
Description: Secondary patency is defined as reestablishment of flow to distal arteries after 100% occlusion has occurred at the target vessel at post-procedure through 6 months.
Time Frame: 6 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 3.7 [1.2 to 8.4]

11. Secondary Outcome: Patency - Primary
Description: Patients were assumed primary patent if the target vessel had continuous flow without revascularization, bypass, or amputation at 9 months.
Time Frame: 9 Months
Population: Intention to Treat (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 95.3 [89.3 to 98.5]

12. Secondary Outcome: Patency - Primary Assisted
Description: Primary assisted patency is defined as continuous flow assisted with a revascularization when the target vessel has restenosed (0-99%) at any time post-procedure through 9 months.
Time Frame: 9 Months
Population: Intention to Treat (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 1.9 [0.2 to 6.6]

13. Secondary Outcome: Patency - Secondary
Description: Secondary patency is defined as reestablishment of flow to distal arteries after 100% occlusion has occurred at the target vessel at post-procedure through 9 months.
Time Frame: 9 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 1.9 [0.2 to 6.6]

14. Secondary Outcome: Target Limb Revascularization
Description: Restenosis is defined as a 50% or greater diameter stenosis observed post-procedure through the 9 month timepoint. Restenosis is initially assessed by Duplex Ultrasound of the iliac artery with the common femoral artery.
Time Frame: 9 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 7.5 [3.6 to 13.3]

15. Secondary Outcome: Restenosis Rate (≥ 50% Diameter Stenosis by Duplex Ultrasound Determination)
Description: as for outcome 14
Time Frame: 9 Months
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 1.9 [0.2 to 6.6]

16. Secondary Outcome: Death
Description: Death can be classified as one of three categories: cardiac, vascular, or non-cardiovascular. All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established.
Time Frame: 9 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 1.5 [0.2 to 5.3]

17. Secondary Outcome: Target Limb Loss
Description: Amputation of the target limb by surgical removal of tissue anywhere from the toe to hip in the ipsilateral limb of the target segment. Amputations are subclassified as: Above the knee, Below the knee, Transmetatarsal, and Toe.
Time Frame: 9 Months
Population: Intention to Treat Population (ITT)
Measure: Number; unit: Percentage of Patients
Arm/Group | Scuba Iliac Stent System
Number analyzed (Participants) | 141
Percentage of Patients | 0 [0 to 1.0]

ADVERSE EVENTS:
Time Frame: From subject index procedure through the 9 month follow-up visit period.
Description: In this study, subjects were encouraged to report adverse events (AEs) spontaneously or in response to general, non-directed questioning (e.g., "How has your health been since the last visit?"). Any time during the study, the subject may volunteer information that resembles an adverse event (AE).
Arm/Group | Scuba Iliac Stent System
Serious Adverse Events (participants affected / at risk) | 47/141
Other Adverse Events (participants affected / at risk) | 35/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scuba Iliac Stent System (N=141)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 3 (3)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 4 (6)
Angina Unstable (Cardiac disorders) | 1 (2)
Atrial Fibrilation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Catheter Site Haemorrhage (General disorders) | 1 (1)
Tenderness (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Post Procedural Infection (Infections and infestations) | 1 (1)
In-stent Arterial Restenosis (Injury, poisoning and procedural complications) | 2 (3)
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 (1)
Stent Occlusion (Injury, poisoning and procedural complications) | 1 (1)
Thrombus in Device (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 1 (1)
Calculus Ureteric (Renal and urinary disorders) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Arterial Thrombus Limb (Vascular disorders) | 1 (2)
Femoral Arterial Stenosis (Vascular disorders) | 3 (3)
Hypertensive Emergency (Vascular disorders) | 1 (1)
Iliac Artery Occlusion (Vascular disorders) | 1 (1)
Iliac Artery Stenosis (Vascular disorders) | 1 (1)
Iliac Artery Thrombosis (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 7 (8)
Leriche Syndrome (Vascular disorders) | 1 (1)
Peripheral Artery Dissection (Vascular disorders) | 1 (2)
Peripheral Embolism (Vascular disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 2 (2)
Subclavian Artery Stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scuba Iliac Stent System (N=141)
Acute Coronary Syndrome (Cardiac disorders) | 3 (3)
Angina Pectoris (Cardiac disorders) | 4 (7)
Catheter Site Haematoma (General disorders) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Femoral Artery Stenosis (Vascular disorders) | 4 (4)
Intermittent Claudication (Vascular disorders) | 9 (13)
Peripheral Artery Dissection (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medtronic has a legitimate interest in ensuring that a multi-center publication is the first publication to be released regarding the completed Study. The Institution agrees that it will not publish or disclose any results of or information pertaining to the study until a multi-center publication is released. If a publication is not released within one year after completion of the study, the Institution will have the right to publish information pertaining to their activities conducted.